CLINICAL TRIAL: NCT03026972
Title: A Phase ⅠStudy of the Human Body Tolerance Research of the Recombinant Mycobacterium Tuberculosis Vaccine Freeze-dried
Brief Title: A Phase ⅠStudy of the Recombinant Mycobacterium Tuberculosis Vaccine Freeze-dried
Acronym: AEC/BC02
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Anhui Zhifei Longcom Biologic Pharmacy Co., Ltd. (Industry)
Collaborators: Shanghai Public Health Clinical Center (Other Government); Beijing Simoonrecord Pharmaceutical Information Consulting Co.,Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: LTao-AEC/BC02-Ⅰ-healthy; LTao (Registry Identifier: AnhuiZhifei)
Record Dates: First submitted 2017-01-12; First posted 2017-01-20 (Estimated); Last update posted 2022-03-24 (Actual); Status verified 2019-12

CONDITIONS: Tuberculosis
Keywords: Safety; Tolerance
MeSH Terms: conditions — Tuberculosis | interventions — Adjuvants, Pharmaceutic; Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Population I (Experimental): Population I has 25 subjects,and it is considered as Tuberculin purified protein derivative(TB-PPD) skin test and specific gamma-interferon (γ-IFN) detection result all negative.Population I are coxal muscle injection of placebo or low dose adjuvant or low dose vaccine.
  Interventions: Biological: Placebo; Biological: Low dose adjuvant; Biological: Low dose vaccine
- Population II (Experimental): Population II is considered as Tuberculin purified protein derivative(TB-PPD) skin test , ESAT6-CFP10 skin test and specific gamma-interferon (γ-IFN) detection result all negative.It has 30 subjects.Population II are coxal muscle injection of placebo or high dose adjuvant or high dose vaccine.
  Interventions: Biological: Placebo; Biological: High dose adjuvant; Biological: High dose vaccine
- Population III (Experimental): Population III is considered as ESAT6-CFP10 skin test and specific gamma-interferon (γ-IFN) detection result negive,but Tuberculin purified protein derivative(TB-PPD) skin test positive.Population IV is needed 30 subjects.These subjects are coxal muscle injection of placebo or high dose adjuvant or high dose vaccine.This arm is uninfected TB PPD positve population.
  Interventions: Biological: Placebo; Biological: High dose adjuvant; Biological: High dose vaccine
- Population IV (Experimental): Population IV is considered as Tuberculin purified protein derivative(TB-PPD) skin test and ESAT6-CFP10 skin test and specific gamma-interferon (γ-IFN) detection result all positive.We are called latent infection population,and need to screen 50 subjects through these three selection method.Population III are coxal muscle injection of placebo or adjuvant( including low dose adjuvant or high dose adjuvant) or vaccine(including low dose vaccine high dose vaccine).
  Interventions: Biological: Placebo; Biological: Low dose adjuvant; Biological: High dose adjuvant; Biological: Low dose vaccine; Biological: High dose vaccine

INTERVENTIONS:
Biological: Placebo — The placebo drug contains 20mg mannitol and 10 millimole(mM) phosphate buffer(PB).population I～population IV are coxal muscle injection of placebo.
Biological: Low dose adjuvant — Population I and polulation IV are coxal muscle injection of low dose adjuvant.
  Arms: Population I; Population IV
Biological: High dose adjuvant — Population II ,Population III and Population IV are coxal muscle injection of high dose adjuvant.
  Arms: Population II; Population III; Population IV
Biological: Low dose vaccine — Population I and population IV are coxal muscle injection of low dose vaccine.
  Arms: Population I; Population IV
Biological: High dose vaccine — Population II,population III and population IV are coxal muscle injection of high dose vaccine .
  Arms: Population II; Population III; Population IV

SUMMARY:
There are four populations in Recombinant Mycobacterium tuberculosis Vaccine Freeze-dried (AEC/BC02) phase I clinical research. The clinical study adopt open research design.

Population I have 25 subjects who received Tuberculin purified protein derivative(TB-PPD) skin test and specific gamma-interferon (γ-IFN)detection whose results are both negative ;Population II have 30 subjects who received Tuberculin purified protein derivative(TB-PPD) and ESAT6-CFP10 skin test in different arms , specific gamma-interferon (γ-IFN) detection whose results are all negative.We call polulation III as uninfected TB PPD positve population.This group screened 30 subjects whose ESAT6-CFP10 skin test and specific gamma-interferon (γ-IFN)detection results are both negative,but Tuberculin purified protein derivative(TB-PPD) skin test positive.50 subjects whose three kinds of detection results are all positive γ-IFN,TB-PPD and ESAT6-CFP10 ) are named as population IV.

After filtrating, injecting of population I start firstly.After ensure the safety of the population I,the population II～polulation IV carry out in turn the implementation at the same time.

DETAILED DESCRIPTION:
Consider the safety of the inoculation,the trial is conducted in the following order:

Population I start firstly, polulation II～population IV is sarted when population I is finished the entire immune and observation safety.Population II and population III should proceed simultaneously,and these two kinds of population finish injecting the first doses of placebo group after 4weeks,population IV start.

All participants of the placebo group and adjuvant group complete the first needle intramuscular injection.5 subjects of Low-dose vaccine group are injected after being sure of the security of placebo and adjucant groups after 3 days. When these low-dose vaccine subjects is sure of safety in 2h,the rest of 5 subjects are injected.Each participant immune one type of placebo, adjuvant or vaccination every two weeks, totally six stitches. In the research, each subject receives only one dose of drug and cannot be subjected to experiments about dose escalation.

The population Ⅰ subjects are received 6 needle times of placebo or low-dose adjuvant or low-dose vaccine by haunch deep intramuscular injection to provide security basis. The subjects should accept some physical examination during the clinical research. Vital signs (breathing, pulse, blood pressure, body temperature) of each volunteer before each needle injection and 30min; and local reaction of each volunteer at 30min after injection;routine blood, routine urine, liver and kidney function, and ECG before first-dose, third-dose,forth-dose and sixth-dose,7 days after the sixth needle injection; Female HCG is tested before each needle injection and 7days after the sixth dose injected; chest X-ray detection before the first injection and 7 days after the sixth needle injection. All subjects should assess the changes of immunological indexes before the first injection, the fourth time before injection and 7 days after the sixth needle injection. The specific injection orders are as follows:

①All the subjects of placebo group(5 cases) and low-dose adjuvant group(10 cases) will be injected on the same day, the adjuvant group subjects should be injected after all the placebo group completed and observed two hours safety;

② All the subjects of low-dose vaccine (10 cases) will be injected on the third day if the placebo group and adjuvant group subjects are observed safety.

③The clinical study of population Ⅱ and population Ⅲ will be carried out 3 days later if the low-dose vaccine group subjects of the population Ⅰ are observed safety; Each subject inoculates a dose of drug every two weeks, a total of six agents. In conclusion, the result of the Phase I Clinical Study of population I evaluate safety of different dose of Recombinant Mycobacterium tuberculosis Vaccine Freeze-dried(AEC/BCO2) in different population, but also provide a safe basis for the Phase I Clinical Study.

The populationⅠsubjects are injected the first needle injection and observe safety after 3 days and then conducted clinical research population Ⅱ and Ⅲ in Phase I Clinical. The study population Ⅱ/Ⅲ will be injected to a placebo or adjuvant or vaccination and collect any adverse events and serious adverse events to evaluate its safety during the period of clinical research.When the above two kinds of population are injected first doses of placebo after 4 weeks,the low-dose group of population IV proceed.High-dose group of population IV conduct trial after the low-dose group injected first dose of placebo later 1 week.

The 30 subjects of study population Ⅱand 30 subjects of population III who meet the inclusion criteria and do not accord with standard of exclusion are divided into placebo group,high-dose adjuvant group and high-dose vaccine group, each group has 10 participants.The 50 subjects of population IV are invidided into low-dose group and high-dose group,each group of 25 subjects.The Low-dose group consiste of 5 placebo subjects,10 adjuvant subjects and 10 vaccine subjects.The high-dose grouping is same as low-dose group.Every subject must accept some physical examination during the clinical research,and all the items of physical examination are as same as population I. Specific injection orders are as follows:

①Population II and population III should proceed simultaneously,and these two kinds of population finish injecting the first doses of placebo group after 4weeks,population IV start;

②High-dose group of population IV conduct trial after the low-dose group injected first dose of placebo later 1 week;

③Every pupolation are injected placebo and adjuvant firstly;5 subjects of Low-dose vaccine group are injected after being sure of the security of placebo and adjucant groups after 3 days. When these low-dose vaccine subjects is sure of safety in 2h,the rest of 5 subjects are injected.

All subjects are vaccinated once every two weeks, a total of six times vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Agreed to participate in the test and sign the informed consent;
* Subjects should comply with the requirements of the clinical trial protocol and be followed;
* Aged form 18-45 years old . Body mass index should be in the range of 18-30. Body Mass Index BMI: weight (Kg)/ [height (m)*height (m)];
* Physical condition: body temperatue, blood pressure, heart rate and respiratory status are normal minor abnormalities but no abnormal symptoms and signs;
* Lab test including blood, urine, liver and kidney function are normal minor abnormalities but no abnormal symptoms and signs;
* ECG,X-ray chest radiograph are normal minor abnormalities but no abnormal symptoms and signs;
* Subjects have no history of tuberculosis;
* Subjects have no acute or chronic disease, acute infectious diseases, dermatoses or skin allergy caused by various reasons;
* Subject have not participated in other clinical drug trials or inoculated against other prophylactic and immune globulin in the nearly 3 months.

Exclusion Criteria:

* Suffering from other serious disease, e.g. tumor, autoimmune disease, progressive atherosclerosis, diabetes accompanied with complications, chronic obstructive pulmonary disease(COPD) needing oxygen therapy, acute or progressive liver or kidney disease, congestive heart failure, etc;
* Subjects were a history of TB;
* Subjects are immune dysfunction or abnormal, e.g. patients receive immunosuppressive agents or immunosuppressive agents, receive immunoglobulin preparations outsider the gastrointestinal or blood products within 3 months, extracted plasma or infected by immunodeficiency virus or related disease;
* Mentally or physically disabled,and have family history of convulsions, epilepsy, encephalopathy or mental illness.
* Subjects have took part in other clinical trials in the nearly 3 months,or vacinated any prophylactic;
* Allergic constitution, e.g. patients have allergic history to two or more kinds of drugs or food, or drug components;
* Substance abuse， drug or alcohol abuse;
* Pregnant or breast feeding female;
* people have birth plan during study or in six moons after entire immune;
* Any other cases that may influence the test evaluation.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2018-09-04 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
The number of participants with Adverse Events after coxal muscle injection | Up to a week after the sixth time injection
  The adverse events observed mainly from laboratory examination(including vital signs/routine blood/routingurine/Liver and kidney fuction/Electrocardiograghy and Chest X-ray detection),skin reactivity and local reaction after drug injection.Vital signs(breathing,pulse,blood pressure,body temperature) of each volunteer before each dose injection,and 30min after injection.Routine blood,routine urine,liver and kidney function,and ECG before first dose,third dose,sixth dose,and 7 days after the sixth time injection;skin reactivity and local reaction of rach volunteer at 30min before and after every injection.

SECONDARY OUTCOMES:
Laboratory markers of immunity | Up to a week after the sixth time injection
  Evaluation of IFN-γand antibody level of before and after the immune,intracellular cytokine staining in blood .

CONTACTS AND LOCATIONS:
Overall Officials: Shuihua Lu, Principal Investigator — Shanghai Public Health Clinical Center
Locations (1):
- Shanghai Public Health clinical Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Young D, Dye C. The development and impact of tuberculosis vaccines. Cell. 2006 Feb 24;124(4):683-7. doi: 10.1016/j.cell.2006.02.013. PMID 16497578
- [Background] Lalvani A, Nagvenkar P, Udwadia Z, Pathan AA, Wilkinson KA, Shastri JS, Ewer K, Hill AV, Mehta A, Rodrigues C. Enumeration of T cells specific for RD1-encoded antigens suggests a high prevalence of latent Mycobacterium tuberculosis infection in healthy urban Indians. J Infect Dis. 2001 Feb 1;183(3):469-77. doi: 10.1086/318081. Epub 2000 Dec 21. PMID 11133379
- [Background] Pathan AA, Wilkinson KA, Klenerman P, McShane H, Davidson RN, Pasvol G, Hill AV, Lalvani A. Direct ex vivo analysis of antigen-specific IFN-gamma-secreting CD4 T cells in Mycobacterium tuberculosis-infected individuals: associations with clinical disease state and effect of treatment. J Immunol. 2001 Nov 1;167(9):5217-25. doi: 10.4049/jimmunol.167.9.5217. PMID 11673535
- [Background] Targeted tuberculin testing and treatment of latent tuberculosis infection. This official statement of the American Thoracic Society was adopted by the ATS Board of Directors, July 1999. This is a Joint Statement of the American Thoracic Society (ATS) and the Centers for Disease Control and Prevention (CDC). This statement was endorsed by the Council of the Infectious Diseases Society of America. (IDSA), September 1999, and the sections of this statement. Am J Respir Crit Care Med. 2000 Apr;161(4 Pt 2):S221-47. doi: 10.1164/ajrccm.161.supplement_3.ats600. No abstract available. PMID 10764341
- [Background] Taylor Z, Nolan CM, Blumberg HM; American Thoracic Society; Centers for Disease Control and Prevention; Infectious Diseases Society of America. Controlling tuberculosis in the United States. Recommendations from the American Thoracic Society, CDC, and the Infectious Diseases Society of America. MMWR Recomm Rep. 2005 Nov 4;54(RR-12):1-81. PMID 16267499
- [Background] Horsburgh CR Jr. Priorities for the treatment of latent tuberculosis infection in the United States. N Engl J Med. 2004 May 13;350(20):2060-7. doi: 10.1056/NEJMsa031667. PMID 15141044
- [Background] Tyagi AK, Nangpal P, Satchidanandam V. Development of vaccines against tuberculosis. Tuberculosis (Edinb). 2011 Sep;91(5):469-78. doi: 10.1016/j.tube.2011.01.003. Epub 2011 Feb 18. PMID 21334259
- [Background] Brandt L, Feino Cunha J, Weinreich Olsen A, Chilima B, Hirsch P, Appelberg R, Andersen P. Failure of the Mycobacterium bovis BCG vaccine: some species of environmental mycobacteria block multiplication of BCG and induction of protective immunity to tuberculosis. Infect Immun. 2002 Feb;70(2):672-8. doi: 10.1128/IAI.70.2.672-678.2002. PMID 11796598
- [Background] McShane H, Hill A. Prime-boost immunisation strategies for tuberculosis. Microbes Infect. 2005 May;7(5-6):962-7. doi: 10.1016/j.micinf.2005.03.009. Epub 2005 Apr 15. PMID 15890555
- [Background] Murray JF. [Current clinical manifestations of tuberculosis]. Rev Prat. 1996 Jun 1;46(11):1344-9. French. PMID 8794617
- [Background] Turner OC, Roberts AD, Frank AA, Phalen SW, McMurray DM, Content J, Denis O, D'Souza S, Tanghe A, Huygen K, Orme IM. Lack of protection in mice and necrotizing bronchointerstitial pneumonia with bronchiolitis in guinea pigs immunized with vaccines directed against the hsp60 molecule of Mycobacterium tuberculosis. Infect Immun. 2000 Jun;68(6):3674-9. doi: 10.1128/IAI.68.6.3674-3679.2000. PMID 10816527
- [Background] Taylor JL, Turner OC, Basaraba RJ, Belisle JT, Huygen K, Orme IM. Pulmonary necrosis resulting from DNA vaccination against tuberculosis. Infect Immun. 2003 Apr;71(4):2192-8. doi: 10.1128/IAI.71.4.2192-2198.2003. PMID 12654841
- [Background] Olsen AW, Williams A, Okkels LM, Hatch G, Andersen P. Protective effect of a tuberculosis subunit vaccine based on a fusion of antigen 85B and ESAT-6 in the aerosol guinea pig model. Infect Immun. 2004 Oct;72(10):6148-50. doi: 10.1128/IAI.72.10.6148-6150.2004. PMID 15385521
- [Background] Andersen P, Doherty TM. TB subunit vaccines--putting the pieces together. Microbes Infect. 2005 May;7(5-6):911-21. doi: 10.1016/j.micinf.2005.03.013. Epub 2005 Apr 14. PMID 15878836
- [Background] Torres M, Herrera T, Villareal H, Rich EA, Sada E. Cytokine profiles for peripheral blood lymphocytes from patients with active pulmonary tuberculosis and healthy household contacts in response to the 30-kilodalton antigen of Mycobacterium tuberculosis. Infect Immun. 1998 Jan;66(1):176-80. doi: 10.1128/IAI.66.1.176-180.1998. PMID 9423855
- [Background] Alexander DC, Liu J. Mycobacteria Genomes. Bacterial Genomes and InfecDis.2003,7(2):153-154.
- [Background] Mostowy S, Cousins D, Brinkman J, Aranaz A, Behr MA. Genomic deletions suggest a phylogeny for the Mycobacterium tuberculosis complex. J Infect Dis. 2002 Jul 1;186(1):74-80. doi: 10.1086/341068. Epub 2002 May 30. PMID 12089664
- [Background] Mostowy S, Onipede A, Gagneux S, Niemann S, Kremer K, Desmond EP, Kato-Maeda M, Behr M. Genomic analysis distinguishes Mycobacterium africanum. J Clin Microbiol. 2004 Aug;42(8):3594-9. doi: 10.1128/JCM.42.8.3594-3599.2004. PMID 15297503
- [Background] Pulendran B, Ahmed R. Immunological mechanisms of vaccination. Nat Immunol. 2011 Jun;12(6):509-17. doi: 10.1038/ni.2039. PMID 21739679
- [Background] Didierlaurent AM, Morel S, Lockman L, Giannini SL, Bisteau M, Carlsen H, Kielland A, Vosters O, Vanderheyde N, Schiavetti F, Larocque D, Van Mechelen M, Garcon N. AS04, an aluminum salt- and TLR4 agonist-based adjuvant system, induces a transient localized innate immune response leading to enhanced adaptive immunity. J Immunol. 2009 Nov 15;183(10):6186-97. doi: 10.4049/jimmunol.0901474. Epub 2009 Oct 28. PMID 19864596
- [Background] He Q, Mitchell A, Morcol T, Bell SJ. Calcium phosphate nanoparticles induce mucosal immunity and protection against herpes simplex virus type 2. Clin Diagn Lab Immunol. 2002 Sep;9(5):1021-4. doi: 10.1128/cdli.9.5.1021-1024.2002. PMID 12204953
- [Background] Vollmer J, Krieg AM. Immunotherapeutic applications of CpG oligodeoxynucleotide TLR9 agonists. Adv Drug Deliv Rev. 2009 Mar 28;61(3):195-204. doi: 10.1016/j.addr.2008.12.008. Epub 2009 Jan 13. PMID 19211030
- [Background] Weeratna RD, McCluskie MJ, Xu Y, Davis HL. CpG DNA induces stronger immune responses with less toxicity than other adjuvants. Vaccine. 2000 Mar 6;18(17):1755-62. doi: 10.1016/s0264-410x(99)00526-5. PMID 10699323
- [Background] Stewart VA, McGrath S, Krieg AM, Larson NS, Angov E, Smith CL, Brewer TG, Heppner DG Jr. Activation of innate immunity in healthy Macaca mulatta macaques by a single subcutaneous dose of GMP CpG 7909: safety data and interferon-inducible protein-10 kinetics for humans and macaques. Clin Vaccine Immunol. 2008 Feb;15(2):221-6. doi: 10.1128/CVI.00420-07. Epub 2007 Dec 12. PMID 18077623
- [Background] Cooper CL, Davis HL, Morris ML, Efler SM, Krieg AM, Li Y, Laframboise C, Al Adhami MJ, Khaliq Y, Seguin I, Cameron DW. Safety and immunogenicity of CPG 7909 injection as an adjuvant to Fluarix influenza vaccine. Vaccine. 2004 Aug 13;22(23-24):3136-43. doi: 10.1016/j.vaccine.2004.01.058. PMID 15297066
- [Background] Halperin SA, Van Nest G, Smith B, Abtahi S, Whiley H, Eiden JJ. A phase I study of the safety and immunogenicity of recombinant hepatitis B surface antigen co-administered with an immunostimulatory phosphorothioate oligonucleotide adjuvant. Vaccine. 2003 Jun 2;21(19-20):2461-7. doi: 10.1016/s0264-410x(03)00045-8. PMID 12744879
- [Background] Jones TR, Obaldia N 3rd, Gramzinski RA, Charoenvit Y, Kolodny N, Kitov S, Davis HL, Krieg AM, Hoffman SL. Synthetic oligodeoxynucleotides containing CpG motifs enhance immunogenicity of a peptide malaria vaccine in Aotus monkeys. Vaccine. 1999 Aug 6;17(23-24):3065-71. doi: 10.1016/s0264-410x(99)00145-0. PMID 10462241
- [Background] Tokunaga T, Yamamoto H, Shimada S, Abe H, Fukuda T, Fujisawa Y, Furutani Y, Yano O, Kataoka T, Sudo T, et al. Antitumor activity of deoxyribonucleic acid fraction from Mycobacterium bovis BCG. I. Isolation, physicochemical characterization, and antitumor activity. J Natl Cancer Inst. 1984 Apr;72(4):955-62. PMID 6200641
- [Background] Krieg AM, Yi AK, Matson S, Waldschmidt TJ, Bishop GA, Teasdale R, Koretzky GA, Klinman DM. CpG motifs in bacterial DNA trigger direct B-cell activation. Nature. 1995 Apr 6;374(6522):546-9. doi: 10.1038/374546a0. PMID 7700380
- [Background] Hornung V, Rothenfusser S, Britsch S, Krug A, Jahrsdorfer B, Giese T, Endres S, Hartmann G. Quantitative expression of toll-like receptor 1-10 mRNA in cellular subsets of human peripheral blood mononuclear cells and sensitivity to CpG oligodeoxynucleotides. J Immunol. 2002 May 1;168(9):4531-7. doi: 10.4049/jimmunol.168.9.4531. PMID 11970999
- [Background] Thomas LJ, Hammond RA, Forsberg EM, Geoghegan-Barek KM, Karalius BH, Marsh HC Jr, Rittershaus CW. Co-administration of a CpG adjuvant (VaxImmune, CPG 7909) with CETP vaccines increased immunogenicity in rabbits and mice. Hum Vaccin. 2009 Feb;5(2):79-84. doi: 10.4161/hv.5.2.6521. Epub 2009 Mar 1. PMID 18670196
- [Background] Chen L, Xu M, Wang ZY, Chen BW, Du WX, Su C, Shen XB, Zhao AH, Dong N, Wang YJ, Wang GZ. The development and preliminary evaluation of a new Mycobacterium tuberculosis vaccine comprising Ag85b, HspX and CFP-10:ESAT-6 fusion protein with CpG DNA and aluminum hydroxide adjuvants. FEMS Immunol Med Microbiol. 2010 Jun 1;59(1):42-52. doi: 10.1111/j.1574-695X.2010.00660.x. Epub 2010 Feb 17. PMID 20298499